CLINICAL TRIAL: NCT00076323
Title: A New Test to Predict the Hemolytic Potential of Drugs in G6PD Deficiency
Brief Title: A Test to Predict the Hemolytic Potential of Drugs in G6PD Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WRAIR 992; G6PD
Record Dates: First submitted 2004-01-20; First posted 2004-01-21 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Glucosephosphate Dehydrogenase Deficiency; Favism
Keywords: G6PD; Favism; G6PD Deficiency; hemolysis; drug reaction; drug-induced hemolysis
MeSH Terms: conditions — Glucosephosphate Dehydrogenase Deficiency; Favism; Hemolysis; Drug-Related Side Effects and Adverse Reactions | interventions — Primaquine

INTERVENTIONS:
Drug: Primaquine

SUMMARY:
This study will evaluate a new and safe testing method for identifying medicines that can cause problems in glucose-6-phosphate dehydrogenase (G6PD) deficient individuals. We are looking for volunteers with G6PD deficiency who would be willing to donate blood samples.

ELIGIBILITY:
Inclusion:

* Normal clinical evaluation
* Willing and able to make all scheduled visits

Exclusion:

* pregnant or planning pregnancy
* Have taken any anti-malarial medication in past month
* Positive blood tests for HIV and specific types of hepatitis
* Allergic to primaquine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14
Dates: Start 2003-12; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Difference in degree of hemolysis of G6PD(-) red blood cells in treated vs untreated matched samples.

CONTACTS AND LOCATIONS:
Overall Officials: Shon A Remich, Principal Investigator — WRAIR, Experimental Therapeutics
Locations (1):
- Walter Reed Army Institute of Research, Silver Spring, Maryland, United States